CLINICAL TRIAL: NCT00091273
Title: Evaluation of Safety and Immunogenicity of a Peptide Vaccine in Patients With Epithelial Ovarian or Primary Peritoneal Cancer
Brief Title: Vaccine Therapy in Treating Patients With Ovarian Epithelial or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Amir Jazaeri, Principal Investigator, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11276; UVACC-OVA3; UVACC-33204
Record Dates: First submitted 2004-09-07; First posted 2004-09-09 (Estimated); Results first posted 2014-06-20 (Estimated); Last update posted 2014-06-20 (Estimated); Status verified 2014-05

CONDITIONS: Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: stage I ovarian epithelial cancer; stage II ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; primary peritoneal cavity cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — incomplete Freund's adjuvant; sargramostim; Chemotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: incomplete Freund's adjuvant
Biological: ovarian cancer peptide vaccine
Biological: sargramostim
Biological: tetanus toxoid helper peptide
Procedure: adjuvant therapy

SUMMARY:
RATIONALE: Vaccines made from peptides may make the body build an immune response to kill tumor cells.

PURPOSE: This phase I trial is studying the side effects of vaccine therapy in treating patients with ovarian epithelial or primary peritoneal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and immunogenicity of adjuvant vaccine comprising ovarian cancer synthetic peptides, tetanus toxoid helper peptide, and sargramostim (GM-CSF) emulsified in Montanide ISA-51 in patients with previously treated ovarian epithelial or primary peritoneal cancer.

OUTLINE: This is an open-label study.

Patients receive vaccine comprising ovarian cancer synthetic peptides, tetanus toxoid helper peptide, sargramostim (GM-CSF), and Montanide ISA-51 subcutaneously and intradermally to 2 different sites on days 1, 8, and 15. On day 22, patients undergo removal of the lymph node draining the vaccination site to determine whether the immune system is responding to the vaccine. Patients then receive additional vaccine as above only to the primary vaccination site on days 29, 36, and 43.

After completion of study treatment, patients are followed at 1 week, 1 month, every 3 months for 9 months, every 6 months for 1 year, and then annually thereafter.

PROJECTED ACCRUAL: A maximum of 9 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed ovarian epithelial or primary peritoneal cancer
* Completed primary therapy (surgery and chemotherapy for newly diagnosed disease) within the past 12 months and meets 1 of the following criteria:

  * Clinical or radiographic evidence of disease
  * Serologic evidence of disease
  * Initial diagnosis of stage III or IV disease AND completed anticancer therapy within the past 12 months
* At least 2 intact axillary and/or inguinal lymph node basins

  * Prior lymph node biopsy allowed provided lymphoscintigraphy demonstrates intact drainage to a node in that basin
* HLA-A1-, -A2-, or -A3-positive

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* GOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count > 1,500/mm^3
* Hemoglobin > 8.0 g/dL OR
* Hematocrit > 25%
* Platelet count ≥ 80,000/mm^3

Hepatic

* AST and ALT ≤ 2.5 times upper limit of normal
* Hepatitis C negative

Renal

* Not specified

Cardiovascular

* No New York Heart Association class III or IV heart disease

Immunologic

* HIV negative
* No active infection requiring antibiotics
* No prior or active autoimmune disorder requiring cytotoxic or immunosuppressive therapy
* No prior autoimmune disorder with visceral involvement
* No known or suspected allergy to any component of the study vaccine
* The following immunologic conditions are allowed:

  * Laboratory evidence of autoimmune disease (e.g., positive antinuclear antibody titer) that is asymptomatic
  * Clinical evidence of vitiligo or other forms of depigmenting illness
  * Mild arthritis requiring non-steroidal anti-inflammatory drugs

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Weight ≥ 110 lbs
* No uncontrolled diabetes, defined as hemoglobin A1C ≥ 7%
* No active hyperthyroidism
* No current or recent (within the past year) addiction to alcohol or drugs
* No medical contraindication or other potential medical problem that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 2 weeks since prior and no concurrent allergy desensitization injections
* More than 2 weeks since prior and no concurrent growth factors (e.g., epoetin alfa or pegfilgrastim)
* More than 1 month since prior and no other concurrent immunotherapy
* More than 2 weeks since prior and no other concurrent potential immunomodulating agents, including any of the following:

  * Interferon
  * Tumor necrosis factor
  * Interleukins or other cytokines
  * Biologic response modifiers
  * Monoclonal antibodies
* No prior vaccination with all of the study peptides relevant to the patient's HLA-type

Chemotherapy

* See Disease Characteristics
* More than 1 month since prior chemotherapy and recovered
* No concurrent cytotoxic chemotherapy

Endocrine therapy

* More than 2 weeks since prior and no concurrent parenteral or oral corticosteroids (e.g., prednisone or albuterol)

  * Topical corticosteroids allowed

Radiotherapy

* More than 1 month since prior radiotherapy and recovered

Surgery

* See Disease Characteristics
* More than 1 month since prior surgery and recovered

Other

* More than 1 month since other prior treatment and recovered
* More than 1 month since prior and no other concurrent investigational agents

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2004-06; Primary Completion 2006-02 (Actual); Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amir A. Jazaeri, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia Cancer Center, Charlottesville, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Arm
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Safety of the Vaccine
Description: Participants kept a toxicity diary during the time frame of interest which was reviewed with a study clinician at each visit.
Time Frame: Days 1,8,15,22,29,36,43,50
Population: All treated subjects were assessed.
Measure: Number; unit: participants
Arm/Group | Single Arm
Number analyzed (Participants) | 9
participants
  # of Subjects Experiencing a DLT | 0
  # of Subjects Not Experiencing a DLT | 9

2. Primary Outcome: Measure of Tumor-antigen-specific Immunity in SIN by ELIspot Assay
Time Frame: Day 22
Population: All treated subjects were assessed.
Measure: Number; unit: participants
Arm/Group | Single Arm
Number analyzed (Participants) | 9
participants
  Responders | 8
  Non-responders | 1

3. Secondary Outcome: Measure of Tumor-antigen-specific Immunity in PBMC by Elispot Assay
Time Frame: Days 1,8,15,22,29,36,43,50 and Month 3
Population: All treated subjects were assessed.
Measure: Number; unit: participants
Arm/Group | Single Arm
Number analyzed (Participants) | 9
participants
  Responders | 8
  Non-responders | 1

ADVERSE EVENTS:
Time Frame: Days 1-50
Arm/Group | Single Arm
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 9/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm (N=9)
Autoimmune Reaction (Immune system disorders) | 2
Hemoglobin (Blood and lymphatic system disorders) | 4
Leukocytes (Blood and lymphatic system disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 2
Fatigue (General disorders) | 7
Fever (General disorders) | 1
Rigors/Chills (General disorders) | 2
Sweating (General disorders) | 2
Bruising (Skin and subcutaneous tissue disorders) | 2
Flushing (Skin and subcutaneous tissue disorders) | 2
Injection Site Reaction (Skin and subcutaneous tissue disorders) | 9
Anorexia (Gastrointestinal disorders) | 1
Dehydration (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Mucositis (Clinical Exam) - Oral Cavity (Gastrointestinal disorders) | 1
Mucositis (Funct/Sympt) - Oral Cavity (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 3
AST (Hepatobiliary disorders) | 2
Alkaline Phosphatase (Hepatobiliary disorders) | 1
Creatinine (Hepatobiliary disorders) | 3
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 3
Hyperkalemia (Metabolism and nutrition disorders) | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Dizziness (Nervous system disorders) | 4
Neuropathy-Sensory (Nervous system disorders) | 1
Pain - Abdomen NOS (General disorders) | 1
Pain - Head/Headache (General disorders) | 6
Pain - Joint (General disorders) | 2
Pain - Muscle (General disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes